CLINICAL TRIAL: NCT05440058
Title: Effect of Timing of Commencement of Bispectral Index Monitoring in Relation to Muscle Relaxant Administration
Brief Title: BIS Monitoring in Relation to Muscle Relaxant Administration
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Matthew J. Ritter, Principal Investigator, Mayo Clinic
Other Study IDs: 22-001485
Record Dates: First submitted 2022-06-27; First posted 2022-06-30 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Cardiovascular Surgery; Bispectral Index; Anesthesia
Keywords: BIS; Paralysis
MeSH Terms: conditions — Paralysis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- BIS Monitoring: Subjects will have BIS sensors applied to forehead
  Interventions: Device: Bispectral Index (BIS) monitoring system

INTERVENTIONS:
Device: Bispectral Index (BIS) monitoring system — Left and right sensors to record EEG activity and muscle reaction to anesthesia utilized in the operating room by anesthesia providers to assess the depth of sedation in patients with anesthesia.

SUMMARY:
The purpose of this study is to determine the overall optimal timing of when the Bispectral Index (BIS) monitor should be started: before or after the muscle relaxant is given.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing elective cardiac surgery
* Muscle relaxation administration by rocuronium

Exclusion Criteria:

* Patient refusal
* Pediatric patients
* Emergency procedure
* Patients with known or suspected carotid or cerebrovascular disease
* Patients with prior stroke
* Skin condition or anatomy preventing proper sensor placement
* Patients who receive ketamine during the study timeframe

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults undergoing elective cardiovascular surgery, for whom BIS monitoring will be used.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2022-08-26 (Actual); Primary Completion 2022-09-20 (Actual); Study Completion 2022-09-20 (Actual)

PRIMARY OUTCOMES:
BIS Values | 25-minute period in the operating room
  Parameters measured from both left and right BIS sensors. BIS monitor algorithm to process EEG information second by second and outputs a number (0-100) that corresponds with a patient's level of consciousness. A level of 0 indicates no EEG activity; a level of 100 indicates awake EEG activity.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Ritter, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials